CLINICAL TRIAL: NCT01371552
Title: Performance Evaluation of a New Daily Disposable Silicone Hydrogel Lens (TUNGSTEN)
Brief Title: Performance Evaluation of a New Daily Disposable Silicone Hydrogel Lens
Acronym: TUNGSTEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P-371-C-100 v2; P/319/08/C (Other: University of Waterloo)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- delefilcon A (Experimental): Part 1: Delefilcon A contact lenses, followed by filcon II 3 contact lenses and narafilcon A contact lenses (in randomized order). Each product worn for three consecutive days, with a minimum 1-day washout between each product. At the conclusion of this wear cycle, the delefilcon A contact lenses were worn in Part 2 for one additional week. All products worn bilaterally in a daily wear, daily disposable modality.
  Interventions: Device: delefilcon A contact lens; Device: filcon II 3 contact lenses; Device: narafilcon A contact lenses
- filcon II 3 (Active Comparator): Part 1: Filcon II 3 contact lenses, followed by narafilcon A contact lenses and delefilcon A contact lenses (in randomized order). Each product worn for three consecutive days, with a minimum 1-day washout between each product. At the conclusion of this wear cycle, the delefilcon A contact lenses were worn in Part 2 for one additional week. All products worn bilaterally in a daily wear, daily disposable modality.
  Interventions: Device: delefilcon A contact lens; Device: filcon II 3 contact lenses; Device: narafilcon A contact lenses
- narafilcon A (Active Comparator): Part 1: Narafilcon A contact lenses, followed by filcon II 3 contact lenses and delefilcon A contact lenses (in randomized order). Each product worn for three consecutive days, with a minimum 1-day washout between each product. At the conclusion of this wear cycle, the delefilcon A contact lenses were worn in Part 2 for one additional week. All products worn bilaterally in a daily wear, daily disposable modality.
  Interventions: Device: delefilcon A contact lens; Device: filcon II 3 contact lenses; Device: narafilcon A contact lenses

INTERVENTIONS:
Device: delefilcon A contact lens — Investigational, silicone hydrogel, single vision contact lens worn on a daily disposable basis for 3 days in Part 1 and one week in Part 2.
Device: filcon II 3 contact lenses — Commercially marketed, silicone hydrogel, single vision contact lens worn on a daily disposable basis for 3 days in Part 1.
  Other Names: Clariti 1-DAY
Device: narafilcon A contact lenses — Commercially marketed, silicone hydrogel, single vision contact lens worn on a daily disposable basis for 3 days in Part 1.
  Other Names: 1-DAY ACUVUE TruEye

SUMMARY:
The purpose of this study was to compare a new daily disposable, silicone hydrogel contact lens to marketed daily disposable, silicone hydrogel contact lenses.

DETAILED DESCRIPTION:
Part 1 of the study involved bilateral wear of three different types of marketed contact lenses. Each type of lens was worn for three consecutive days of daily disposable wear. Participants had been previously identified as symptomatic lens wearers or asymptomatic lens wearers, based upon their responses to a screening questionnaire. Participants wore each lens type for as long as they were comfortable during the day, but lenses were removed before sleep. After completion of Part 1, participants began Part 2, which included dispensing of the investigational study lens for up to one week of bilateral wear, with a single follow-up visit at the end of that period.

ELIGIBILITY:
Inclusion Criteria:

* 17 years of age; full legal capacity to volunteer.
* Ocular examination within the last two years
* Correctable to a visual acuity of 20/30 or better (in each eye) with habitual vision correction.
* Currently wearing soft contact lenses.
* Clear corneas; no active ocular disease.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Currently wearing 1-DAY ACUVUE TruEye or Sauflon Clariti 1-DAY contact lenses.
* Monovision.
* Any ocular disease.
* Never worn contact lenses before.
* Corneal refractive surgery.
* Uses topical ocular medicine.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FAAO, Principal Investigator — Centre for Contact Lens Research, School of Optometry, University of Waterloo
Locations (1):
- University of Waterloo Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center in Canada.
Pre-assignment Details: 10 people were enrolled but not dispensed into Part 1 due to failing inclusion/exclusion criteria.
Groups:
- Delefilcon A / Filcon II 3 / Narafilcon A: Part 1: Delefilcon A, then Filcon II 3, then Narafilcon A, 3 days each. Part 2: Delefilcon A for 1 week.
- Narafilcon A / Filcon II 3 / Delefilcon A: Part 1: Narafilcon A, then Filcon II 3, then Delefilcon A, 3 days each. Part 2: Delefilcon A for 1 week.
- Filcon II 3 / Narafilcon A / Delefilcon A: Part 1: Filcon II 3, then Narafilcon A, the Delefilcon A, 3 days each. Part 2: Delefilcon A for 1 week.
- Delefilcon A / Narafilcon A / Filcon II 3: Part 1: Delefilcon A, then Narafilcon A, then Filcon II 3, 3 days each. Part 2: Delefilcon A for 1 week.
- Narafilcon A / Delefilcon A / Filcon II 3: Part 1: Narafilcon A, then Delefilcon A, then Filcon II 3, 3 days each. Part 2: Delefilcon A for 1 week.
- Filcon II 3 / Delefilcon A / Narafilcon A: Part 1: Filcon II 3, then Delefilcon A, then Narafilcon A, 3 days each. Part 2: Delefilcon A for 1 week.
Period: Part 1, First 3 Days
Arm/Group | Delefilcon A / Filcon II 3 / Narafilcon A | Narafilcon A / Filcon II 3 / Delefilcon A | Filcon II 3 / Narafilcon A / Delefilcon A | Delefilcon A / Narafilcon A / Filcon II 3 | Narafilcon A / Delefilcon A / Filcon II 3 | Filcon II 3 / Delefilcon A / Narafilcon A
Started | 19 | 17 | 20 | 20 | 15 | 18
Completed | 19 | 17 | 19 | 20 | 15 | 18
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Inconvenience | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 1, Second 3 Days
Arm/Group | Delefilcon A / Filcon II 3 / Narafilcon A | Narafilcon A / Filcon II 3 / Delefilcon A | Filcon II 3 / Narafilcon A / Delefilcon A | Delefilcon A / Narafilcon A / Filcon II 3 | Narafilcon A / Delefilcon A / Filcon II 3 | Filcon II 3 / Delefilcon A / Narafilcon A
Started | 19 | 17 | 18 (1 subject discontinued after First 3 days due to positive slit lamp findings unrelated to lens wear) | 20 | 15 | 18
Completed | 18 (One subject did not complete period due to discomfort but continued to next, as allowed by protocol) | 17 | 18 | 20 | 15 | 18
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Third 3 Days
Arm/Group | Delefilcon A / Filcon II 3 / Narafilcon A | Narafilcon A / Filcon II 3 / Delefilcon A | Filcon II 3 / Narafilcon A / Delefilcon A | Delefilcon A / Narafilcon A / Filcon II 3 | Narafilcon A / Delefilcon A / Filcon II 3 | Filcon II 3 / Delefilcon A / Narafilcon A
Started | 19 | 17 | 18 | 20 | 15 | 18
Completed | 19 | 17 | 18 | 20 | 14 (One subject did not complete period due to randomization error, but continued into Part 2.) | 17 (One subject did not complete period due to discomfort, but continued into Part 2.)
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Period: Part 2, One Week
Arm/Group | Delefilcon A / Filcon II 3 / Narafilcon A | Narafilcon A / Filcon II 3 / Delefilcon A | Filcon II 3 / Narafilcon A / Delefilcon A | Delefilcon A / Narafilcon A / Filcon II 3 | Narafilcon A / Delefilcon A / Filcon II 3 | Filcon II 3 / Delefilcon A / Narafilcon A
Started | 18 (One participant discontinued between Part 1 and Part 2 due to inconvenience) | 17 | 18 | 20 | 15 | 18
Completed | 18 | 17 | 18 | 20 | 15 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This reporting group includes all enrolled participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 119
Age Continuous [Mean (Standard Deviation); unit: years] | 27 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 30
Region of Enrollment [Number; unit: participants]
  Canada | 119

OUTCOME MEASURES:

1. Primary Outcome: Mean Value of Comfort During the Day
Description: The participant recorded a number from 0 to 100 in response to the question, "How would you rate the comfort of your lenses over the last hour?" in which 0 = very poor and 100 = excellent. Comfort was assessed at 4 hours, 8 hours, and 12 hours, and the responses were averaged.
Time Frame: Part 1: Day 2 at 4 hours, 8 hours, and 12 hours
Population: This reporting group includes all participants who completed 12 hours of lens wear on Day 2.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Delefilcon A: Delefilcon A contact lenses worn in a daily disposable mode for 3 days in Part 1
- Filcon II 3: Filcon II 3 contact lenses worn in a daily disposable mode for 3 days in Part 1
- Narafilcon A: Narafilcon A contact lenses worn in a daily disposable mode for 3 days in Part 1
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 94 | 88 | 85
Units on a scale | 89 (11) | 85 (13) | 86 (13)

2. Primary Outcome: Mean Overall Comfort Given at End of Wear
Description: The participant recorded a number from 0 to 100 in response to the question, "How would you rate the overall comfort of these lenses?" in which 0 = very poor and 100 = excellent. The end of wear questionnaire was completed at time of lens removal for that day.
Time Frame: Part 1: Day 3
Population: This reporting group includes all participants who completed all three lens wear periods in Part 1.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 104 | 104 | 104
Units on a scale | 90 (10) | 83 (16) | 86 (15)

3. Primary Outcome: Mean Overall Quality of Vision at End of Wear
Description: The participant recorded a number from 0 to 100 in response to the question, "How would you rate the overall quality of vision while wearing these lenses?" in which 0 = very poor and 100 = excellent. The end of wear questionnaire was completed at time of lens removal for that day.
Time Frame: Part 1: Day 3
Population: This reporting group includes all participants who completed all three lens wear periods in Part 1.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 104 | 104 | 104
Units on a scale | 91 (10) | 87 (12) | 88 (13)

4. Primary Outcome: Mean Overall Ease of Handling at End of Wear
Description: The participant recorded a number from 0 to 100 in response to the question, "How would you rate the overall ease of handling these lenses?" in which 0 = very difficult and 100 = very easy. The end of wear questionnaire was completed at time of lens removal for that day.
Time Frame: Part 1: Day 3
Population: This reporting group includes all participants who completed all three lens wear periods in Part 1.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 104 | 104 | 104
Units on a scale | 90 (13) | 91 (12) | 93 (10)

5. Primary Outcome: Percentage of Participants Reporting That Their Eyes Rarely or Never Felt Dry at End of Wear
Description: The participant circled a number from 0 to 4 in response to the question, "Over the entire day while wearing these contact lenses, how often did your eyes feel dry?" in which 0 = never, 1 = rarely, 2 = sometimes, 3 = frequently, 4 = constantly. The end of wear questionnaire was completed at time of lens removal for that day.
Time Frame: Part 1: Day 2
Population: This reporting group includes all participants who completed all three lens wear periods in Part 1.
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 104 | 104 | 104
Percentage of participants | 63 | 38 | 57

6. Primary Outcome: Percentage of Participants Preferring Study Lens Either Strongly or Slightly (of Those With a Preference) vs. Their Habitual Lenses at End of Wear
Description: The participant circled a number from 1 to 5 in response to the question, "Overall, which lens do you prefer - the lens you wore today or your regular lenses?" in which 1 = strongly prefer my regular lenses, 2 = prefer my regular lenses, 3 = no preference, 4 = prefer test lens, 5 = strongly prefer test lens. The end of wear questionnaire was completed at time of lens removal for that day.
Time Frame: Part 1: Day 3
Population: This reporting group includes all participants who completed all three lens wear periods in Part 1.
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 104 | 104 | 104
Percentage of participants | 62 | 35 | 54

7. Primary Outcome: Lens Wettability
Description: Lens wettability was assessed by the investigator during slit-lamp examination and graded on a 0-4 scale in 0.25 steps, where 0 = excellent and 4 = severely reduced.
Time Frame: Part 1: Day 1 at Dispense, Day 1 at 8 hours, Day 3 at 8 hours
Population: This reporting group includes all participants who completed all three lens wear periods in Part 1.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Number analyzed (Participants) | 104 | 104 | 104
Units on a scale
  Day 1 at Dispense | 0.25 (0.39) | 0.49 (0.50) | 0.46 (0.46)
  Day 1 at 8 hours | 0.46 (0.50) | 0.77 (0.55) | 0.89 (0.69)
  Day 3 at 8 hours | 0.51 (0.47) | 0.76 (0.66) | 0.91 (0.72)

8. Primary Outcome: Percentage of Participants Responding "Yes"
Description: The participant responded to 11 subjective, performance-related statements on a questionnaire by circling 1 = yes, 2 = no, or 3 = don't know.
Time Frame: Part 2: Day 7
Population: This reporting group includes all participants who completed Part 2.
Measure: Number; unit: Percentage of participants
Groups:
- Delefilcon A - All Wearers: Delefilcon A contact lenses worn in a daily disposable mode for 7 days in Part 2, all wearers
Arm/Group | Delefilcon A - All Wearers
Number analyzed (Participants) | 106
Percentage of participants
  These lenses provide excellent comfort | 85
  These lenses provide excellent quality of vision | 87
  These lenses are very easy to handle | 83
  These lenses are very easy to insert on my eye | 88
  Lenses provide excellent comfort during the day | 89
  Lenses provide excellent comfort at the end of day | 64
  So comfortable I almost forget I am wearing lenses | 67
  Deliver comfort/vision long days/demanding schedul | 72
  Total package-great vision, comfort, convenience | 73
  My life is demanding. Lenses meet those demands | 64
  I need high performance-these lenses deliver | 70

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: The safety reporting group includes all enrolled and exposed participants.
Arm/Group | Delefilcon A | Filcon II 3 | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/117 | 0/117
Other Adverse Events (participants affected / at risk) | 0/117 | 12/117 | 1/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Delefilcon A (N=117) | Filcon II 3 (N=117) | Narafilcon A (N=117)
Redness (Eye disorders) | 0/115 | 12 | 1/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.